CLINICAL TRIAL: NCT04186169
Title: Preliminary Studies to Evaluate the Impact of Peri-Atrial Inflammatory Fat Tissue on Atrial Fibrillation Using Ultra-High Resolution CT
Brief Title: Peri-Atrial Inflammatory Fat and Atrial Fibrillation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left the institution
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00210289
Record Dates: First submitted 2019-12-02; First posted 2019-12-04 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Intervention Model Description: Arm 1: Paroxysmal AF (n=100). Observational. Arm 2: Persistent AF (n=50). PVI arm Arm 3: Persistent AF (n=50). PVI + fat-targeted ablation arm
Who Masked: Participant
Masking Description: Neither the patients nor the operators are NOT blinded as to whether the patients receive the ultra-high resolution CT or the standard CT. For patients with paroxysmal AF, there is no blinding because there is only one group. The patients with persistent AF will be blinded as to whether they are assigned to the PVI group or the PVI + Fat ablation group. The operators are not blinded (single-blinded design).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm 1: Paroxysmal AF - PVI arm (Placebo Comparator): The subjects with paroxysmal AF undergo pulmonary vein isolation (PVI).
  Interventions: Procedure: Catheter ablation
- Arm 2: Persistent AF - PVI arm (Placebo Comparator): The subjects with persistent AF undergo pulmonary vein isolation (PVI).
  Interventions: Procedure: Catheter ablation
- Arm 3: Persistent AF - PVI + Fat-targeted ablation (Experimental): The subjects with persistent AF undergo pulmonary vein isolation (PVI) and additional ablation to target the inflammatory fat tissue
  Interventions: Procedure: Catheter ablation

INTERVENTIONS:
Procedure: Catheter ablation — Catheter ablation

SUMMARY:
Atrial fibrillation (AF) impacts the lives of 30 million people worldwide. Pulmonary vein isolation (PVI) by catheter ablation is effective for paroxysmal AF, but the success rate remains marginal at 60-80%. For persistent AF, defined as continuous AF that sustains longer than 7 days, the success rate is even lower. The low success rate of AF ablation reflects the fact that there is no effective target identified to modify the underlying substrate beyond PVI. Recently, investigators have made an exciting discovery that higher mean CT attenuation values of peri-atrial fat tissue, correlated with inflammatory fat, are associated with higher incidence of recurrence after AF ablation. In this protocol, investigators will investigate the clinical significance of peri-atrial inflammatory fat tissue in AF using ultra-high resolution CT.

DETAILED DESCRIPTION:
Investigators will prospectively enroll 200 adult participants referred to the Johns Hopkins Hospital for catheter ablation of atrial fibrillation (AF). Investigators will first enroll participants with paroxysmal AF (n=100) to complete sensitivity analysis of inflammatory fat and potential target identification before enrolling participants with persistent AF (n=100). All participants (n=200) will undergo pre-procedural CT using the ultra-high resolution CT scanner 3-4 days prior the ablation procedure to allow a sufficient amount of time for image processing. In all participants (n=200), blood specimens will be collected immediately prior to the ablation procedure. The participants with paroxysmal AF (n=100) will receive the standard of care, which is PVI, and the clinical outcome will be followed up to 12 months post-procedure. In this group, investigators will conduct a sensitivity analysis to define the range of peri-left atrial (LA) fat tissue (in HU) that is associated with AF recurrence. Investigators will also conduct computation of source-sink mismatch arising from wall thinning due to fat infiltration into the myocardium that favors functional block and local reentry. For participants with persistent AF (n=100), investigators will conduct an exploratory clinical trial where the participants will be randomly assigned to 1) PVI group (n=50), or 2) PVI + inflammatory fat-targeted ablation group (n=50). In the latter group, additional focal ablation will be performed beyond PVI to target the inflammatory fat tissue based on the result of the sensitivity analysis. Randomization will be performed with the use of an automated computer-generated randomization algorithm. The participants will be unaware of the group assignment, but the operators will not be blinded (single-blinded design). In all patients, no ablation strategies beyond PVI except cavotricuspid isthmus (CTI) ablation for typical atrial flutter (AFL) will be allowed, such as linear lesions (e.g. roof lines, mitral isthmus lines), and focal ablation to eliminate complex fractionated atrial electrograms (CFAE) and rotating drivers.

ELIGIBILITY:
Inclusion criteria:

* Ages 18 to 100 years
* Adult men and women undergoing the first catheter ablation of AF for whom cardiac CT is clinically indicated to guide the procedure.

Exclusion criteria:

* Inability to provide consent
* Estimated glomerular filtration rate (eGFR) <30 mL/min/1.73 m^2
* Known history of anaphylaxis to radiocontrast

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-02-19 (Actual); Primary Completion 2024-11-12 (Actual); Study Completion 2024-11-12 (Actual)

PRIMARY OUTCOMES:
Freedom from any documented episode of AF | 12 months
  Freedom from any documented episode of AF lasting longer than 30 seconds after the performance of a single ablation procedure without the use of antiarrhythmic drugs (AADs). No episode of AF occurring within the initial 3-month blanking period after ablation will be counted. An episode of AF will be considered part of the primary outcome analyses if it lasts longer than 30 seconds and is documented by any form of monitoring, regardless of symptoms. A repeat left atrial (LA) ablation procedure at any time will also be considered to constitute a recurrence for the purpose of the outcome analyses. Participants who complete fewer than 3 months of follow-up and thus do not complete the blanking period will be excluded from endpoint analysis. There will be no blanking period after a second procedure.

SECONDARY OUTCOMES:
Freedom from documented AF after two ablation procedures | 12 months
  Freedom from documented AF after two ablation procedures
Freedom from any documented atrial arrhythmia after one ablation procedure | 12 months
  Freedom from any documented atrial arrhythmia after one ablation procedure
Freedom from any documented atrial arrhythmia after two ablation procedures | 12 months
  Freedom from any documented atrial arrhythmia after two ablation procedures
Use of antiarrhythmia drugs (AADs) | 12 months
  Use of antiarrhythmia drugs (AADs) will be measured as a categorical variable (Yes or No).
Procedure time | 12 months
  Procedure time will be measured as a continuous variable (in minutes).
Occurrence of repeat procedures | 12 months
  Occurrence of repeat procedures will be measured as a categorical variable (Yes or No).
Occurrence of peri-procedural complications | 30 days
  Occurrence of peri-procedural complications will be measured as a categorical variable (Yes or No).

CONTACTS AND LOCATIONS:
Overall Officials: Hiroshi Ashikaga, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ciuffo L, Nguyen H, Marques MD, Aronis KN, Sivasambu B, de Vasconcelos HD, Tao S, Spragg DD, Marine JE, Berger RD, Lima JAC, Calkins H, Ashikaga H. Periatrial Fat Quality Predicts Atrial Fibrillation Ablation Outcome. Circ Cardiovasc Imaging. 2019 Jun;12(6):e008764. doi: 10.1161/CIRCIMAGING.118.008764. Epub 2019 Jun 10. PMID 31177816